CLINICAL TRIAL: NCT00406796
Title: FVF3565s Intravitreal Ranibizumab (rhuFab V2) in the Treatment of Macular Edema Associated With Perfused Central (CRVO) Retinal Venous Occlusive Disease
Brief Title: Lucentis for Central Retinal Vein Occlusion (CRVO)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: California Retina Consultants (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Dante J Pieramici, California Retina Consultants and Research Foundation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FVF3565s
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Central Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 0.5mg Ranibizumab
  Interventions: Drug: Ranibizumab
- 2 (Active Comparator): 0.3mg Ranibizumab
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 0.3mg and 0.5mg dose of Ranibizumab 0.05ml administered intravitreally
  Other Names: Lucentis

SUMMARY:
The purpose of this study is to determine whether ranibizumab will be effective in reducing if not eliminating the macular edema associated with the disease, central retinal vein occlusion (CRVO).

DETAILED DESCRIPTION:
Retinal Venous Occlusive disease is the second only to diabetic retinopathy as a major cause of blindness associated with retinal vascular disease. Macular edema is a major cause of vision loss in patients presenting with central abd hemi vein occlusions. Currently, there is no proven treatment to address macular edema in these patients. In the past laser photocoagulation has been used, but was found to offer no visual benefits over the natural history in the treatment of macular edema associated with CRVO. Investigators have demonstrated in case reports that intravitreal triamcinolone (Kenalog) may result in the reduction in macular edema, leading to visual improvement in some patients with CRVO. Triamcinolone is relatively well tolerated in many patients, but its use is associated with significant risk of elevated intraocular pressure, cataract, and intraocular infection.

Ranibizumab (rhuFab V2, an anti-VEGF agent, is a potent inhibitor of vascular permeability, with the potential to reduce retinal vascular leakage and diminish macular edema. In addition, as an anti-VEGF agent, it may also inhibit neovascularization of the iris, a frequent complication of ischemic central retinal vein occlusion. Ranibizumab use as an intravitreal agent does carry the risk of intraocular infection but probably carries very low risk of glaucoma or cataract formation, making it a potentially safer pharmacologic treatment for CRVO associated macular edema as compared to triamcinolone

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Clinical evidence of perfused central retinal vein occlusion. A central retinal vein occlusion (CRVO) is defined as an eye that has retinal hemorrhages and a dilated retinal venous system in all 4 quadrants. Other evidence of a CRVO may include telangiectatic capillary bed and collateral vessels at the optic nerve head.
* Central macular edema present on clinical examination and OCT testing with a central point thickness > 250 microns
* Visual acuity score greater than or equal to 19 letters (20/400) and less than or equal to 73 letters (20/40) by the ETDRS visual acuity protocol.
* Media clarity, pupillary dilation and patient cooperation sufficient to allow OCT testing and retinal photography

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or known to be pregnant, also premenopausal women not using adequate contraception.
* Participation in another simultaneous ocular investigation or trial
* Patient with uncontrolled hypertension
* Patient has a condition that, in the opinion of the investigator would preclude participation in the study (i.e. chronic alcoholism, drug abuse)
* Patient has significant diabetic retinopathy (greater than moderate NPDR) or macular edema associated with diabetic retinopathy
* Exam or OCT reveals evidence of vitreoretinal interface abnormality that may be contributing to the macular edema
* Eye that in the investigator has no chance of improvement in visual acuity following resolution of macular edema (i.e subretinal fibrosis or geographic atrophy)
* Presence of another ocular condition that may affect the visual acuity or macular edema during the course of the study (i.e AMD, uveitis, Irvine-Gas)
* Evidence of neovascularization of the iris or retina (presence of ischemic CRVO)
* Presence of substantial cataract, one that might decrease the vision by 3 or more lines of vision at sometime during the study.
* History of Grid/Focal laser or Panretinal laser in the study eye
* History of vitreous surgery in the study eye
* History of use of intravitreal, peribulbar, or retrobulbar steroids within six months of the study.
* History of Cataract Surgery within 6 months of enrollment.
* History of YAG capsulotomy within 2 months of the surgery.
* Visual acuity <20/400 in the fellow eye
* Uncontrolled Glaucoma, pressure >30 despite treatment with glaucoma medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2008-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the proportion of subjects in each group ( 0.3, 0.5 mg ) gaining 15 or more letters at month 6 and 12 (ETDRS visual refraction at 4 meters) and to determine if a difference exists between the high and low dose. | 6 and 12 months

SECONDARY OUTCOMES:
To determine the safety and tolerability of ranibizumab in the treatment of macular edema associated with CRVO in each group | 6 and 12 months
To determine the proportion of subjects in each group gaining 15 or more letters at month 3, 6, 9 & 12 as compared to baseline (ETDRS visual refraction at 4 meters) and to determine if a statistically significant difference exists between the groups | 3, 6, 9, and 12 months
Change in central retinal thickness from baseline as measured by OCT at months 3, 6, 9 and 12 | 3,6,9, and 12 months
To determine the proportion of subjects in each group losing 15 or more letters at months 3,6,9,12 as compared to baseline (ETDRS visual refraction at 4 meters) and to determine if a statistically significant difference exists between the groups. | 3, 6, 9, and 12 months
To determine the proportion of subjects in each group losing 30 or more letters at months 3,6,8,12 as compared to baseline (ETDRS visual refraction at 4 meters) and to determine if a statistically significant difference exists between the groups. | 3, 6, 9, and 12 months
To determine if changes in best-corrected visual acuity are correlated with changes in total macular volume, center point thickness, and/or central 1mm subfield thickness. | Months 1-12

CONTACTS AND LOCATIONS:
Overall Officials: Dante J Pieramici, M.D., Principal Investigator — California Retina Consultants
Locations (4):
- United States (4):
  - California Retina Consultants, Bakersfield, California
  - California Retina Consultants, Oxnard, California
  - California Retina Consultants, Santa Barbara, California
  - California Retina Consultants, Santa Maria, California